CLINICAL TRIAL: NCT03911141
Title: Behavioral Economic Approaches to Increase Physical Activity Among Patients With Elevated Risk for Cardiovascular Disease
Acronym: BE ACTIVE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: 831230
Record Dates: First submitted 2019-04-03; First posted 2019-04-10 (Actual); Results first posted 2025-01-27 (Actual); Last update posted 2025-01-27 (Actual); Status verified 2024-12

CONDITIONS: Atherosclerotic Cardiovascular Disease
MeSH Terms: conditions — Atherosclerosis

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Control (No Intervention): Participants receive a daily text message stating whether or not they achieved their step goal on the prior day during the 12 months of intervention and 6 months of follow-up.
- Gamification Intervention (Experimental): Participants have an 8-week ramp-up period where daily goals increase from baseline to the step target, and sign a pledge agreeing to try their best to meet their goals.
  Participants are entered into a game. Each week they receive 70 points. Each day they're told their step count and points. If the step goal was met they keep their points, but if not, they lose 10 points. At the end of the week if they have at least 40 points they move up a level, but if not, they drop a level. Participants start in the middle of 5 levels.
  Participants choose a support partner who gets a weekly email with the participant's progress. We hold a 3-way phone call with the participant and supportive sponsor to discuss ways they can help the participant meet their goal. Every 8 weeks, have a follow up call if the participant is stuck in a lower level and restart them back at the middle level.
  In the follow-up period, participants continue to get a daily text stating if they met their step goal.
  Interventions: Behavioral: Gamification
- Financial Incentive Intervention (Experimental): Participants are informed that each week that money is placed in a virtual account for them. Each day the participant is informed of their step count on the prior day. If the step goal was achieved, the balance remains. Each day the goal is not achieved, the participant is informed that some of the money was taken away. We will use an 8-week ramp-up period in which daily goals are increased gradually from baseline to targets.
  During the follow-up period, participants in this arm will continue to receive a daily text message stating whether or not they achieved their step goal on the prior day.
  Interventions: Behavioral: Financial
- Gamification and Financial Incentive Intervention (Experimental): Participants receive both of the interventions described in the Gamification Intervention arm and the Financial Incentive Intervention arm.
  Interventions: Behavioral: Gamification; Behavioral: Financial

INTERVENTIONS:
Behavioral: Gamification — Participants have an 8-week ramp-up period where daily goals increase from baseline to the step target, and sign a pledge agreeing to try their best to meet their goals.
  Participants are entered into a game. Each week they receive 70 points. Each day they're told their step count and points. If the step goal was met they keep their points, but if not, they lose 10 points. At the end of the week if they have at least 40 points they move up a level, but if not, they drop a level. Participants start in the middle of 5 levels.
  Participants choose a support partner who gets a weekly email with the participant's progress. We hold a 3-way phone call with the participant and supportive sponsor to discuss ways they can help the participant meet their goal. Every 8 weeks, have a follow up call if the participant is stuck in a lower level and restart them back at the middle level.
  In the follow-up period, participants continue to get a daily text stating if they met their step goal.
  Arms: Gamification Intervention; Gamification and Financial Incentive Intervention
Behavioral: Financial — Participants are informed that each week money is placed in a virtual account for them. Each day the participant is informed of their step count on the prior day. If the step goal was achieved, the balance remains. Each day the goal is not achieved, the participant is informed that some of the money was taken away. We will use an 8-week ramp-up period in which daily goals are increased gradually from baseline to targets.
  During the follow-up period, participants in this arm will continue to receive a daily text message stating whether or not they achieved their step goal on the prior day.
  Arms: Financial Incentive Intervention; Gamification and Financial Incentive Intervention

SUMMARY:
The objective of this study is to use a randomized, controlled trial to test the effectiveness of using gamification, financial incentives, or both to increase physical activity among patients with elevated risk for atherosclerotic cardiovascular disease (ASCVD). ASCVD is the leading cause of morbidity and mortality in the United States. Regular physical activity has been shown to reduce the risk of ASCVD, but less than 50% of US adults achieve enough physical activity to obtain these benefits.

DETAILED DESCRIPTION:
Atherosclerotic cardiovascular disease (ASCVD) is the leading cause of morbidity and mortality in the United States (US). Regular physical activity has been demonstrated to reduce the risk of ASCVD and is associated with a number of other health benefits. Yet, less than 50% of adults in the US achieve enough physical activity to actually obtain these benefits. Insights from behavioral economics have been shown to both better reflect the 'predictable irrationality' of humans and to be effective in designing interventions that achieve sustained improvements in health behavior. Our prior work has demonstrated that interventions using financial incentives and gamification can leverage principles from behavioral economics to increase physical activity during 3-month interventions and sustain effects in 3-month follow-up periods. These findings warrant further investigation of longer-term effects. In this study, we conduct a four-arm randomized, controlled trial to evaluate the effectiveness of using behavioral economic approaches including gamification, financial incentives, or both to increase physical activity among patients with elevated risk for atherosclerotic cardiovascular disease during a 12-month intervention with a 6-month follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* Have a 10-year ASCVD risk score of 7.5% or greater (including those with existing ASCVD)
* Are able to provide informed consent

Exclusion Criteria:

* Are already participating in another physical activity study
* An 18-month physical activity program is infeasible (e.g. metastatic cancer; unable to ambulate or provide informed consent) or unsafe (currently pregnant or told by a physician not to exercise)
* They do not have a device (e.g. smartphone, tablet, or computer) to transmit data from the wearable activity tracker
* Baseline step count is 7,500 or greater
* They do not have a primary care physician in the University of Pennsylvania Health System.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1062 (Actual)
Dates: Start 2019-04-12 (Actual); Primary Completion 2023-07-24 (Actual); Study Completion 2024-01-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mitesh Patel, MD, MBA, MS, Principal Investigator — University of Pennsylvania; Alexander Fanaroff, MD, MHS, Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Derived] Russell LB, Volpp KGM, Patel MS, Chokshi NP, Coratti S, Farraday D, Norton L, Rareshide C, Zhu J, Klaiman T, Szymczak JE, Small DS, Fanaroff AC. Cost-Effectiveness of Gamification, Financial Incentives, or Both to Increase Physical Activity Among Patients With Elevated Risk for Cardiovascular Disease. Circ Cardiovasc Qual Outcomes. 2025 Jul;18(7):e011839. doi: 10.1161/CIRCOUTCOMES.124.011839. Epub 2025 Jun 17. PMID 40525292
- [Derived] Ryu E, Farraday D, Fanaroff AC, Coratti S, Chokshi NP, Zhu J, Szymczak JE, Russell LB, Norton L, Small D, Volpp KG, Klaiman T. What motivates participants: a qualitative analysis of gamification and financial incentives to increase physical activity. BMC Public Health. 2025 May 16;25(1):1804. doi: 10.1186/s12889-025-22717-0. PMID 40380122
- [Derived] Fanaroff AC, Patel MS, Chokshi N, Coratti S, Farraday D, Norton L, Rareshide C, Zhu J, Klaiman T, Szymczak JE, Russell LB, Small DS, Volpp KGM. Effect of Gamification, Financial Incentives, or Both to Increase Physical Activity Among Patients at High Risk of Cardiovascular Events: The BE ACTIVE Randomized Controlled Trial. Circulation. 2024 May 21;149(21):1639-1649. doi: 10.1161/CIRCULATIONAHA.124.069531. Epub 2024 Apr 7. PMID 38583084
- [Derived] Fanaroff AC, Patel MS, Chokshi N, Coratti S, Farraday D, Norton L, Rareshide C, Zhu J, Szymczak JE, Russell LB, Small DS, Volpp KGM. A randomized controlled trial of gamification, financial incentives, or both to increase physical activity among patients with elevated risk for cardiovascular disease: rationale and design of the be active study. Am Heart J. 2023 Jun;260:82-89. doi: 10.1016/j.ahj.2023.02.014. Epub 2023 Mar 2. PMID 36870551

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Before randomization, participants completed a baseline period where they wore a Fitbit for two weeks for the study team to track their average daily step counts. Week two of the baseline period was used to determine eligibility. The average of step counts over 1000 steps per day were taken to calculate the baseline step count. Participants with baseline steps over 7,500 were considered ineligible.
Groups:
- Financial Incentive Intervention: Participants are informed that each week that money is placed in a virtual account for them. Each day the participant is informed of their step count on the prior day. If the step goal was achieved, the balance remains. Each day the goal is not achieved, the participant is informed that some of the money was taken away. We will use an 8-week ramp-up period in which daily goals are increased gradually from baseline to targets.
  During the follow-up period, participants in this arm will continue to receive a daily text message stating whether or not they achieved their step goal on the prior day.
  Financial: Participants are informed that each week money is placed in a virtual account for them. Each day the participant is informed of their step count on the prior day. If the step goal was achieved, the balance remains. Each day the goal is not achieved, the participant is informed that some of the money was taken away. We will use an 8-week ramp-up period in which daily goals are increased gradually from baseline to targets.
  During the follow-up period, participants in this arm will continue to receive a daily text message stating whether or not they achieved their step goal on the prior day.
Period: Overall Study
Arm/Group | Control | Gamification Intervention | Financial Incentive Intervention | Gamification and Financial Incentive Intervention
Started | 151 | 304 | 302 | 305
Completed | 144 | 263 | 286 | 280
Not Completed | 7 | 41 | 16 | 25

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control | Gamification Intervention | Financial Incentive Intervention | Gamification and Financial Incentive Intervention | Total
Number analyzed (Participants) | 151 | 304 | 302 | 305 | 1062
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.6 (8) | 67.2 (8) | 66.4 (8.2) | 66.6 (8.2) | 66.7 (8.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 97 | 197 | 173 | 175 | 642
  Male | 54 | 107 | 129 | 130 | 420
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White non-Hispanic | 103 | 214 | 202 | 218 | 737
  Black non-Hispanic | 40 | 76 | 82 | 68 | 266
  Asian non-Hispanic | 7 | 5 | 7 | 9 | 28
  Hispanic | 1 | 4 | 7 | 4 | 16
  Other | 0 | 5 | 4 | 6 | 15
Education [Count of Participants; unit: Participants]
  Some high school | 2 | 1 | 3 | 4 | 10
  High school graduate | 13 | 14 | 19 | 6 | 52
  Some college or specialized training | 31 | 69 | 57 | 58 | 215
  College graduate | 105 | 220 | 223 | 237 | 785
Marital Status [Count of Participants; unit: Participants]
  Single | 27 | 48 | 40 | 44 | 159
  Married | 91 | 189 | 189 | 195 | 664
  Other | 33 | 67 | 73 | 66 | 239
Annual Household Income [Count of Participants; unit: Participants]
  Less than $50,000 | 48 | 61 | 73 | 61 | 243
  $50,000 to $100,000 | 52 | 109 | 106 | 106 | 373
  Greater than $100,000 | 51 | 134 | 123 | 138 | 446
Self reported health status [Count of Participants; unit: Participants]
  Excellent | 11 | 23 | 11 | 21 | 66
  Very Good | 56 | 96 | 95 | 88 | 335
  Good | 60 | 145 | 149 | 147 | 501
  Fair | 23 | 37 | 45 | 47 | 152
  Poor | 1 | 3 | 2 | 2 | 8
Prior wearable device use [Count of Participants; unit: Participants] | 106 | 213 | 206 | 214 | 739
BMI [Mean (Standard Deviation); unit: kg/m^2] | 31.4 (7.3) | 31 (6.3) | 31.5 (7) | 31.1 (6.5) | 31.2 (6.7)
Diabetes [Count of Participants; unit: Participants] | 37 | 65 | 66 | 76 | 244
Hyperlipidemia [Count of Participants; unit: Participants] | 77 | 163 | 170 | 155 | 565
Hypertension [Count of Participants; unit: Participants] | 93 | 188 | 192 | 184 | 657
Current smoking [Count of Participants; unit: Participants] | 11 | 10 | 11 | 11 | 43
Prior myocardial infarction [Count of Participants; unit: Participants] | 4 | 6 | 8 | 7 | 25
Stroke [Count of Participants; unit: Participants] | 2 | 4 | 7 | 5 | 18
Heart Failure [Count of Participants; unit: Participants] | 4 | 6 | 5 | 5 | 20
Chronic obstructive pulmonary disease [Count of Participants; unit: Participants] | 5 | 4 | 10 | 9 | 28
Chronic kidney disease [Count of Participants; unit: Participants] | 4 | 8 | 10 | 15 | 37
Baseline daily steps [Mean (Standard Deviation); unit: Average daily step counts] | 4980 (1554) | 4958 (1556) | 5018 (1579) | 5081 (1585) | 5014 (1569)
Step goal selection [Count of Participants; unit: Participants]
  33% increase from baseline | 51 | 92 | 95 | 114 | 352
  40% increase from baseline | 26 | 37 | 45 | 56 | 164
  50% increase from baseline | 21 | 72 | 61 | 55 | 209
  Custom goal | 53 | 103 | 101 | 80 | 337
Step goal increase from baseline [Mean (Standard Deviation); unit: step counts] | 1855 (867) | 1890 (854) | 1890 (829) | 1826 (742) | 1867 (817)

OUTCOME MEASURES:

1. Primary Outcome: Change in Mean Daily Step Counts During the 12 Month Intervention Using a Wearable Pedometer (Fitbit Watch) to Measure Step Count.
Description: Change in mean daily steps counts from baseline to the 12-month intervention period, excluding the 8-week ramp-up phase. This will be measured using the Fitbit Charge wearable device.
Time Frame: Months 1-12
Measure: Mean (Standard Deviation); unit: Step counts
Arm/Group | Control | Gamification Intervention | Financial Incentive Intervention | Gamification and Financial Incentive Intervention
Number analyzed (Participants) | 151 | 304 | 302 | 305
Step counts | 1418 (1753) | 1954 (1706) | 1915 (1903) | 2297 (1842)

2. Secondary Outcome: Change in Mean Daily Step Counts During the 6 Month Follow-up Using a Wearable Pedometer (Fitbit Watch) to Measure Step Count.
Description: Change in mean daily steps from baseline to the post-intervention follow-up period. This will be measured using the Fitbit Charge wearable device.
Time Frame: Months 1-18
Measure: Mean (Standard Deviation); unit: Step counts
Arm/Group | Control | Gamification Intervention | Financial Incentive Intervention | Gamification and Financial Incentive Intervention
Number analyzed (Participants) | 151 | 304 | 302 | 305
Step counts | 1245 (1879) | 1708 (1882) | 1576 (2062) | 1831 (1891)

3. Secondary Outcome: Change in Mean Daily Minutes of Moderate to Vigorous Physical Activity (MVPA) During the 12 Month Intervention Using a Wearable Device (Fitbit Watch) to Measure MVPA Derived From Step Counts.
Description: Change in mean daily minutes of MVPA from baseline to the intervention period, excluding the 8-week ramp up phase. This will be measured using the Fitbit Charge wearable device.
Time Frame: Months 1-12
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | Control | Gamification Intervention | Financial Incentive Intervention | Gamification and Financial Incentive Intervention
Number analyzed (Participants) | 151 | 304 | 302 | 305
Minutes | 5.3 (9.5) | 7.4 (10.6) | 7.8 (11.1) | 9 (10.5)

4. Secondary Outcome: Change in Mean Daily Minutes of Moderate to Vigorous Physical Activity (MVPA) During the 6 Month Follow-up Using a Wearable Device (Fitbit Watch) to Measure MVPA Derived From Step Counts.
Description: Change in mean daily minutes of MVPA from baseline to the post-intervention follow-up period. This will be measured using the Fitbit Charge wearable device.
Time Frame: Months 1-18
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | Control | Gamification Intervention | Financial Incentive Intervention | Gamification and Financial Incentive Intervention
Number analyzed (Participants) | 151 | 304 | 302 | 305
Minutes | 4.7 (10.2) | 5.4 (11.2) | 5.3 (10.9) | 5.5 (10.4)

5. Other Pre Specified Outcome: Proportion of Weeks That Achieve 150 Minutes of MVPA During the 12 Month Intervention Using a Wearable Device (Fitbit Watch) to Measure MVPA Derived From Step Counts.
Description: Proportion of weeks that achieve at least 150 minutes of MVPA per week from baseline to the intervention period. The denominator is the total number of weeks all participants in each arm participated in the study and the numerator is the number of weeks all participants had at least 150 minutes of MVPA. This will be measured using the Fitbit Charge wearable device.
Time Frame: Months 1-12
Measure: Number; unit: Proportion of weeks
Arm/Group | Control | Gamification Intervention | Financial Incentive Intervention | Gamification and Financial Incentive Intervention
Number analyzed (Participants) | 151 | 304 | 302 | 305
Proportion of weeks | .16 | .23 | .24 | .27

6. Other Pre Specified Outcome: Proportion of Weeks That Achieve 150 Minutes of MVPA During the 6 Month Follow-up Using a Wearable Device (Fitbit Watch) to Measure MVPA Derived From Step Counts.
Description: Proportion of weeks that achieve at least 150 minutes of MVPA per week from baseline to the follow-up period. The denominator is the total number of weeks all participants in each arm participated in the study and the numerator is the number of weeks all participants had at least 150 minutes of MVPA. This will be measured using the Fitbit Charge wearable device.
Time Frame: Months 1-18
Measure: Number; unit: Proportion of weeks
Arm/Group | Control | Gamification Intervention | Financial Incentive Intervention | Gamification and Financial Incentive Intervention
Number analyzed (Participants) | 151 | 304 | 302 | 305
Proportion of weeks | .14 | .18 | .18 | .20

ADVERSE EVENTS:
Time Frame: 18 months
Description: Adverse events were collected via participant report through study surveys at 6-months, 12-months and 18 months or participant report to study staff through text, email or phone call.
Arm/Group | Control | Gamification Intervention | Financial Incentive Intervention | Gamification and Financial Incentive Intervention
All-Cause Mortality (participants affected / at risk) | 0/151 | 1/304 | 0/302 | 0/305
Serious Adverse Events (participants affected / at risk) | 21/151 | 51/304 | 45/302 | 44/305
Other Adverse Events (participants affected / at risk) | 80/151 | 180/304 | 140/302 | 171/305
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Control (N=151) | Gamification Intervention (N=304) | Financial Incentive Intervention (N=302) | Gamification and Financial Incentive Intervention (N=305)
Orthopedic (Musculoskeletal and connective tissue disorders) | 8 (8) | 12 (12) | 11 (12) | 14 (16)
Cardiovascular (Cardiac disorders) | 2 (2) | 9 (11) | 11 (16) | 5 (6)
Fitbit-related (Product Issues) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Other (General disorders) | 11 (11) | 33 (37) | 26 (33) | 25 (33)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Control (N=151) | Gamification Intervention (N=304) | Financial Incentive Intervention (N=302) | Gamification and Financial Incentive Intervention (N=305)
Orthopedic (Musculoskeletal and connective tissue disorders) | 35 (49) | 86 (106) | 55 (69) | 81 (98)
Cardiovascular (Cardiac disorders) | 4 (4) | 9 (11) | 15 (21) | 9 (10)
Fitbit-related (Product Issues) | 4 (4) | 4 (6) | 5 (6) | 8 (8)
Other (General disorders) | 37 (52) | 85 (124) | 66 (92) | 73 (110)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-05-30): https://cdn.clinicaltrials.gov/large-docs/41/NCT03911141/Prot_SAP_000.pdf